CLINICAL TRIAL: NCT03563547
Title: Effects of a Fat Modified Diet Enriched With Soy Protein on Cholesterol Levels in Children Affected With Heterozygous Familial Hypercholesterolemia: a Randomized Controlled Study
Brief Title: Effects of Soy Protein on Cholesterol Levels in Children Affected With Familial Hypercholesterolemia
Acronym: SOYFIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Austrian Academic Institute for Clinical Nutrition (Other)
Collaborators: Medical University of Vienna (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SoyfitKW01
Record Dates: First submitted 2018-06-11; First posted 2018-06-20 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Heterozygous Familial Hypercholesterolemia
Keywords: LDL-Cholesterol; Heterozygous Familial Hypercholesterolemia; Paediatrics; Dietary Treatment
MeSH Terms: interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fat modified diet (Active Comparator): Subjects in this arm had been instructed to achieve specific daily maximum intakes in total fat (≤ 30% of total energy intake), saturated fatty acids (≤10% of total fat intake) and cholesterol (≤ 300 mg). Furthermore the participating families had been trained to replace as many visible fat sources as possible with rapeseed oil due to its favorable composition of polyunsaturated fatty acids.
  Interventions: Behavioral: Dietary counseling (fat modifed diet)
- Fat modifed diet enriched with soy protein (Experimental): Subjects in this arm had been instructed to achieve specific daily maximum intakes in total fat (≤ 30% of total energy intake), saturated fatty acids (≤10% of total fat intake) and cholesterol (≤ 300 mg). Furthermore the participating families had been trained to replace as many visible fat sources as possible with rapeseed oil due to its favorable composition of polyunsaturated fatty acids.
  Subjects in this arm were additionally instructed to consume at least 0.25 g of soy protein per kg bodyweight per day and were provided with recipes and practical advice on how to achieve this goal. Example provided: a child with a bodyweight of 30kg would have to consume the equivalent of approx. 50g of Tofu per day to meet the treatment target.
  Interventions: Behavioral: Dietary Counseling (fat modified + soy enriched diet)

INTERVENTIONS:
Behavioral: Dietary counseling (fat modifed diet) — Subjects in both groups had been instructed to achieve specific daily maximum intakes in total fat (≤ 30% of total energy intake), saturated fatty acids (≤10% of total fat intake) and cholesterol (≤ 300 mg). Furthermore the participating families had been trained to replace as many visible fat sources as possible with rapeseed oil due to its favorable composition of polyunsaturated fatty acids.
  Arms: Fat modified diet
Behavioral: Dietary Counseling (fat modified + soy enriched diet) — Subjects in both groups had been instructed to achieve specific daily maximum intakes in total fat (≤ 30% of total energy intake), saturated fatty acids (≤10% of total fat intake) and cholesterol (≤ 300 mg). Furthermore the participating families had been trained to replace as many visible fat sources as possible with rapeseed oil due to its favorable composition of polyunsaturated fatty acids.
  Subjects allocated to the soy group and their families were additionally instructed to consume at least 0.25 g of soy protein per kg bodyweight per day and were provided with recipes and practical advice on how to achieve this goal. Example provided: a child with a bodyweight of 30kg would have to consume the equivalent of approx. 50g of Tofu per day to meet the treatment target.
  Arms: Fat modifed diet enriched with soy protein

SUMMARY:
Familial hypercholesterolemia (FH) is an inheritable, autosomal dominant disorder leading to pathologically increased levels of low-density-lipoprotein cholesterol (LDL-C). Dietary treatment remains an important tool in the management of affected children even after the decision for the initiation of pharmacotherapy is made. However, little evidence is available on the beneficial effects of diets low in saturated fat and cholesterol and diets enriched with soy in children affected with FH. Based on these previous findings we hypothesize that the LDL-C lowering effect of a fat-modified diet could be further increased by the addition of soy-protein in children affected with HeFH.

DETAILED DESCRIPTION:
This study is a prospective randomized controlled trial. The enrolled subjects were recruited from the outpatient clinic for disorders of metabolism of the Medical University of Vienna. Subjects were either allocated into a group treated with a dietary regimen high in unsaturated fats, low in saturated fats and enriched with soy-protein ("soy group") or a group treated with a diet high in unsaturated fats and low in saturated fats ("control group") alone at random. All subjects had been instructed to adhere to a fat-modified diet as described below prior to enrolment into the study as part of their routine treatment. Prior to being considered for inclusion in the study all subjects had to undergo nutritional protocoling using 24h dietary recall protocols, which were completed by their legal guardians, for 7 days. This was done to confirm adherence to the routine dietary treatment. Furthermore, all patients had been screened for metabolic diseases other than FH as part of their initial routine assessment in our specialised centre.

Subjects in both groups had been instructed to achieve specific daily maximum intakes in total fat (≤ 30% of total energy intake), saturated fatty acids (≤10% of total fat intake) and cholesterol (≤ 300 mg). Furthermore the participating families had been trained to replace as many visible fat sources as possible with rapeseed oil due to its favorable composition of polyunsaturated fatty acids.24 Subjects allocated to the soy group and their families were additionally instructed to consume at least 0.25 g of soy protein per kg bodyweight per day and were provided with recipes and practical advice on how to achieve this goal. Example provided: a child with a bodyweight of 30kg would have to consume the equivalent of approx. 50g of Tofu per day to meet the treatment target. This dosage had been reported as effective for LDL-C reduction in children in a previous, non-controlled study.10

Further appointments with an experienced dietitian were made after enrolment for both treatment groups, totalling 7 training sessions (60 minutes each) over the course of the first 7 weeks of the trial. This was done to identify possible issues with the practical implementation of especially the soy-enriched diet.

Patients were asked to provide weekly urine samples and blood was drawn immediately after enrolment, week 7 and week 13, respectively. The urine- and plasma samples were immediately frozen and later analysed for their isoflavone content. Isoflavone levels were assessed at baseline to verify that the respective patients did not consume soy products prior to the trial. All enrolled subjects had to participate for 13 weeks or were excluded from the statistical evaluation (per protocol analysis). If relevant levels of isoflavones were detected in either urine or plasma of subjects in the Control-group the subjects were to be excluded from any further statistical evaluation.

The study was approved by the Ethics Committee of the Medical University of Vienna. Informed consent from all participating subjects and their legal guardians was obtained prior to their enrolment in the study. Our research was conducted in accordance with the latest Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent of both the patient and their legal guardian, age of 4 to 14, diagnosis of definite FH using the Simon Broome criteria, body weight within normal age-specific percentile range (Kromeyer-Hauschild et al.), the proven ability and willingness to adhere to a fat-modified diet.

Exclusion Criteria:

* Metabolic or genetic disorders other than FH, current infectious disease, current or history of cancerous disease, current treatment with lipid lowering drugs, failure to complete all trial-related assessments, reported habit of consuming soy products or adherence to a non-standard diet (e.g. vegetarianism) prior to enrolment into the study.

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2009-09-03 (Actual); Primary Completion 2014-10-09 (Actual); Study Completion 2017-10-09 (Actual)

PRIMARY OUTCOMES:
LDL-C change from baseline | 13 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Austrian Academic Institute for Clinical Nutrition, Vienna, Austria

REFERENCES:
- [Derived] Helk O, Widhalm K. Effects of a low-fat dietary regimen enriched with soy in children affected with heterozygous familial hypercholesterolemia. Clin Nutr ESPEN. 2020 Apr;36:150-156. doi: 10.1016/j.clnesp.2019.09.009. Epub 2020 Jan 31. PMID 32220359